CLINICAL TRIAL: NCT01517425
Title: Evaluating Cardiovascular Phenotypes Using Induced Pluripotent Stem Cells
Acronym: iPSC
Status: Enrolling by invitation | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute, Scripps Translational Science Institute
Other Study IDs: 11-5676
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Subjects previously enrolled in the Scripps Genebank Study
- Controls: Subjects previously enrolled in the Scripps Healthy Elderly Active Longevity (HEAL) Cohort

SUMMARY:
This research is being done to understand how changes in DNA may put people at risk for developing coronary artery disease. Stem cells will be made using cells from blood and/or skin biopsy samples. We are trying to understand which specific changes in DNA negatively impact a person's health.

ELIGIBILITY:
Inclusion Criteria:

Cases:

1. Previously enrolled in the CAD module of the Genebank at Scripps Clinic Registry
2. Eligible to have their blood drawn
3. Be reliable, cooperative and willing to comply with all protocol-specified procedures
4. Able to understand and grant informed consent

Controls:

1. Previously enrolled in the Healthy Elderly Active Longevity (HEAL) Cohort
2. Eligible to have their blood drawn
3. Be reliable, cooperative and willing to comply with all protocol-specified procedures
4. Able to understand and grant informed consent

Exclusion Criteria:

1. Unwilling or unable to grant informed consent.
2. Have a significant medical condition that in the Investigator's opinion may interfere with subject's study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects previously enrolled in the Scripps Genebank or Healthy Elderly Active Longevity (HEAL) Cohort
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-11; Primary Completion 2025-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
iPSC development | five years
  Develop methods of iPSC generation from patients with genomic risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States